CLINICAL TRIAL: NCT04663178
Title: The Effect of Warm Salt Water Foot Bath on the Management of Chemotherapy Induced Fatigue
Brief Title: Foot Bath and Chemotherapy Induced Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ferda AKYUZ OZDEMIR, MsCN, The Effect of Warm Salt Water Foot Bath on the Management of Chemotherapy Induced Fatigue, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Warm Salt Water Foot Bath
Record Dates: First submitted 2020-12-02; First posted 2020-12-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapeutic Toxicity; Chemotherapy-induced Fatigue
Keywords: Chemotherapy Induced Fatigue; Warm salt water foot bath

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Salt Water Foot Bath Group (Experimental): In the first interview Patient Identification Form, Fatigue Severity and Piper Fatigue Scale (PFS) were applied to the patients. A training booklet about chemotherapy-induced fatigue containing the definition, causes, ad development process of chemotherapy-induced fatigue and effective coping approaches were delivered to patients.
  Each patient received iodine salt and a liquid thermometer to measure the temperature of the water. The patients were asked 1 day after the treatment to apply warm salt water bath of 41-42ºC once a day for 20 minutes for 7 days.
  Subsequently, the fatigue level of the patients was evaluated 30 minutes after having a warm saltwater foot bath and recorded by questioning via calling them with phone every day and using the Visual Fatigue Scale for 7 days. In the last interview PFS was used to evaluate the effect level of fatigue on the quality of life and the assessment process was completed.
  Interventions: Other: Warm Salt Water Foot Bath
- Control Group (No Intervention): A training booklet about chemotherapy-induced fatigue
  In the first interview Patient Identification Form, Fatigue Severity and Piper Fatigue Scale were applied to the patients.
  A training booklet about chemotherapy-induced fatigue containing the definition, causes, ad development process of chemotherapy-induced fatigue and effective coping approaches were delivered to experimental group.
  Subsequently, the fatigue level of the patients was evaluated and recorded by questioning via calling them with phone every day and using the Visual Fatigue Scale for 7 days. The patients were evaluated in the evening. In the last interview conducted with the patient on the 7th day, Piper's Fatigue Scale was used to evaluate the effect level of fatigue on the quality of life and the assessment process was completed.

INTERVENTIONS:
Other: Warm Salt Water Foot Bath — A training booklet about chemotherapy-induced fatigue + 20-minute warm salt water application to their feet for a week after the treatment by explaining and showing the video prepared about the preparation and practice of warm salt water foot bath.
  Arms: Warm Salt Water Foot Bath Group

SUMMARY:
Background: In a limited number of studies conducted with the participation of cancer patients, it has been reported that warm water bath may be beneficial for management of cancer-related fatigue.

Objective: This experimental study was conducted to evaluate the effect of warm salt water foot bath applied to reduce the chemotherapy-induced fatigue.

Interventions/Methods: Seventy-nine patients who were experiencing moderate or higher level of fatigue were included in this study conducted between November 2017-February 2018. 42 of the patients were assigned to the experimental group and 37 patients were assigned to the control group. A training booklet about chemotherapy-induced fatigue were given to all patients. In addition, the experimental group was asked to perform 20-minute warm salt water application to their feet for a week after the treatment by explaining and showing the video prepared about the preparation and practice of warm salt water foot bath. Subsequently, the patients were called by phone every day for one week to record their fatigue levels.

Results: The 7-day fatigue course of both groups was similar. However the physical, emotional, affective and cognitive distress related to fatigue decreased in the experimental group but did not decrease in the control group.

Conclusion: The warm salt water footbath may be an effective approach in enhancing fatigue related quality of life. However, it is needed to conduct more comprehensive studies to express the effectiveness.

Implications to Practice: Nurses can propose the use of the warm salt water footbath in the management of chemotherapy induced fatigue.

Keywords: Chemotherapy Induced Fatigue, Warm salt water foot bath

DETAILED DESCRIPTION:
Cancer is an important health problem that is seen frequently in the society and causes a large number of people to lose their lives today. Turkey Statistics Institute's report stating that 81.129 people living in Turkey lost their lives in 2018 due to cancer has further increased the importance of this issue.

The main treatment approaches used in the treatment of cancer are surgical treatment, chemotherapy, and radiotherapy. Being one of these treatment approaches, chemotherapy causes many side effects such as low blood count, fatigue, alopecia, change in taste/smell, nausea-vomiting, mucositis, constipation, diarrhoea, loss of appetite, and neuropathy and adversely affects the quality of life and compliance to treatment. Fatigue, which is one of these problems, is one of the main problems that is frequently reported by patients and adversely affects the daily activities of patients. The incidence of fatigue in patients undergoing chemotherapy has been reported to be 82-96%. Many studies have reported that 30% of patients continue to experience fatigue feeling even in the post-treatment period. Many patients have expressed that they have difficulty in performing activities of daily living and experience difficulty in focusing, lack of strength, apathy towards activities, mood disorders, and loss of sexual desire due to fatigue. Therefore, extensive examination and management of fatigue are important to ensure the compliance to treatment in these patients, increase the treatment efficacy, and enhance their quality of lives.

In the literature, the use of many pharmacological and non-pharmacological approaches in the management of chemotherapy-induced fatigue is recommended. While pharmacological approaches such as methylphenidate, modafinil, and erythrocyte transfusion ensure patients to cope with fatigue by generally treating the problems causing the development of fatigue, non-pharmacological approaches such as training of the patients as well as their families, increasing activity level, yoga, Tai-Chi and Reiki practice, cognitive behavioural therapy approach, energy saving, nutrition regulation, music therapy and massage strengthen patients and support them to cope with fatigue.

This experimental study was conducted in the Outpatient Chemotherapy Unit of the Institute of Oncology in Istanbul University between 15 November 2017 and 28 February 2018 after obtaining institutional permission and ethics committee approval. After giving information about the study, the patients who agreed to participate in the study were divided into experimental (n = 38) or control (n = 37) groups using a randomisation list prepared by random number method in Excel program by the researcher. Interactive training and training booklet containing the definition, causes, ad development process of chemotherapy-induced fatigue and effective coping approaches were delivered to both groups. In addition; in order to cope with chemotherapy-induced fatigue, the experimental group patients were asked 1 day after the treatment to apply warm salt water bath of 41-42ºC once a day for 20 minutes between 21:00-22:00 at home for 7 days and when chemotherapy related fatigue was at the highest level. By using 10-minute video previously prepared by the researcher, how the patient will prepare and apply the temperature of the warm salt water of 41-42oC and the salt rate (280 grams of table salt to 8 litres of water) to be used for footbath were shown and explained.

ELIGIBILITY:
Inclusion Criteria:

* Receiving adjuvant or neoadjuvant chemotherapy with the diagnosis of early stage cancer
* Having fatigue severity of 3 and >3
* Agreeing to participate in the study.

Exclusion Criteria:

* Having the complaint of peripheral neuropathy.
* Being diagnosed with diabetes
* Having impaired skin integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Patient Identification Form | One week
  This form, which was prepared by the researcher in accordance with the literature and consisting of seven sections, contains 29 questions evaluating the personal characteristics of the patients, the characteristics of the disease and the treatment process, and the functional adequacy of the patient.
Fatigue Severity | One week
  The severity of fatigue was classified depending on NCI-CTCAE v3.0 adverse events classification system for fatigue: "0" for "I am not tired", "1" for "I am slightly tired, relieved by rest"; "2" for "I am moderately tired, not relieved by rest"; "3" for "I am very tired, not relieved by rest and is limited instrumental activities of daily living", "4" for "I am extremely tired", fatigue is not relieved by rest and is limited self-care activities of daily living.
Piper Fatigue Scale | One week
  The questions the fatigue-related behavioural, affective, sensory and cognitive distress level of the patients in 22 items and 4 subscales. In each item of the scale, emotions that may be felt due to fatigue are ranged from 1 (weak) to 10 (strong). The person defines his/her fatigue he/she experiences at that moment by marking the best answer (number) reflecting it. Fatigue-related subscale scores (behavioural, affective, sensory and cognitive) are obtained by summing the scores of all items in that subscale and dividing the resulting score to number of items. The overall fatigue score is obtained by summing the score of all items and dividing them by the total number of items. The subscale and general scale score ranges from 0 to 10 and the increased score indicates increased perceived fatigue. There are also 5 open-ended questions in the scale and these questions are not included in the score calculation of fatigue perception.

CONTACTS AND LOCATIONS:
Overall Officials: Ferda AKYUZ OZDEMIR, Principal Investigator — IUC Florence Nıghtingale Nursing Faculty
Locations (1):
- Outpatient Chemotherapy Unit of the Institute of Oncology in Istanbul University, Istanbul, Sisli, Turkey (Türkiye)